CLINICAL TRIAL: NCT05232968
Title: Ameliorating Effects of Aging by Physical Exercise: Molecular, Metabolic and Structural Adaptations, Multi-organ Integrative Approach
Brief Title: Ameliorating Effects of Aging by Physical Exercise
Acronym: AMETHYST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Ukropcová, MD, PhD, Professor, Slovak Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APVV-20-0466
Record Dates: First submitted 2022-01-14; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Aging; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elderly volunteers participating in the long-term exercise program (Experimental): Elderly volunteers will be recruited from participants in the long-term exercise program (ongoing since 2017) at the Center of Physical Activity BMC SAS in Bratislava.
  Interventions: Other: Long-term exercise program
- Elderly sedentary volunteers (No Intervention): Control population will be recruited from the sedentary elderly, who dropped out from the exercise program ≥2 years prior entering this study and do not exercise on regular basis.
- Elderly volunteers participating in the short-term exercise program (Experimental): Elderly volunteers will follow 4-month of aerobic-strength training intervention and exercise induced effects on mild cognitive impairment will be determined afterwards.
  Interventions: Other: Short-term exercise program

INTERVENTIONS:
Other: Long-term exercise program — Training intervention (aerobic-strength training) will combine a 1-hour aerobics training, which requires movement coordination, and two 1-hour lessons, combining strength load (25 minutes, 50-60% 1RM, which gradually increases in proportion to increasing strength, 8-12 repetitions, training all major muscle groups) and aerobic exercise (25 minutes of Nordic walking or stationary bike), with a short warm-up at the beginning and stretching at the end. The individualized training program will be based on the determination of physical fitness (Rockport gait test) and muscle strength (dynamometry).
  Arms: Elderly volunteers participating in the long-term exercise program
Other: Short-term exercise program — Training intervention (aerobic-strength training) will combine a 1-hour aerobics training, which requires movement coordination, and two 1-hour lessons, combining strength load (25 minutes, 50-60% 1RM, which gradually increases in proportion to increasing strength, 8-12 repetitions, training all major muscle groups) and aerobic exercise (25 minutes of Nordic walking or stationary bike), with a short warm-up at the beginning and stretching at the end. The individualized training program will be based on the determination of physical fitness (Rockport gait test) and muscle strength (dynamometry).
  Arms: Elderly volunteers participating in the short-term exercise program

SUMMARY:
With increasing longevity, a significant increase in the incidence of neurodegenerative diseases is expected. According to forecasts based on data from the World Health Organization and data from epidemiological studies, up to 106 million people will have Alzheimer's disease in 2050, it's 1 in 85 people living on the planet. If it will be possible to manage to delay the onset or slow the progression of the disease by a single year, it will mean 9.2 million fewer patients worldwide. This leaves considerable scope for options to modify the onset and prevalence of the disease through lifestyle changes such as eating habits and exercise. It is known that the human brain retains a certain natural plasticity even in old age, which is a great advantage that allows it to adapt to physiological stimuli, such as regular exercise. The pleiotropic beneficial effects of exercise therefore have considerable potential to be used in the prevention and slowing of the progression of cognitive and motor function decline as well as in the prevention / treatment of metabolic dysregulation. This fact is supported by many epidemiological and interventional studies with exercise, emphasizing the importance of the global trend to use exercise as a standardized method of prevention and treatment of many chronic diseases and cognitive deficits.

DETAILED DESCRIPTION:
This interventional study will examine the effects of a comprehensive intervention associated with regular short-term (4 months) and long-term (≥2 years) exercise on the cognitive and motor functions of patients with mild cognitive impairment, as well as the effect of aging, physical activity profile and physical fitness on physiological functions (metabolism, motor skills, cognition) and bioactive molecules.

The study will be carried out in the Department of Internal Medicine and in the Center for Physical Activity Research of the Biomedical Center of the Slovak Academy of Sciences in Bratislava.

Recruitment and screening of seniors with MCI will be carried out by psychologists from the Memory Center in Bratislava (http://www.centrummemory.sk/) and neurologists from II. Department of Neurology LFUK and UNB. All volunteers will be informed in detail about the objectives of the study, the examinations and study protocol, the benefits as well as the potential risks associated with its completion and will sign an informed consent. The study protocol is approved by the ethics committee of the Bratislava.

The project aims to study the effects and mechanisms of the positive impact of regular physical activity and increased physical fitness on health and processes associated with aging, with emphasis on metabolic, cognitive and motor functions, physical fitness and bioactive molecules in the circulation and skeletal muscle. It therefore has real potential to reveal new physiologically important mechanisms, biomarkers or even potential molecular targets for the therapy of neurodegenerative and metabolic diseases. One of the important goals of the project is the implementation of the obtained results into clinical practice, in cooperation with clinicians, psychologists, trainers and special educators.

ELIGIBILITY:
Inclusion Criteria:

* 55-85 years of age,
* non-smokers
* complete vaccination against COVID19
* continuation in the supervised exercise program (for study of long-term effects of exercise experimental group)
* sedentary lifestyle ≥2 years prior this study (for group without intervention),
* mild cognitive impairment (for study of short-term effects of exercise experimental group)
* absence of any psychological, sociological or geographical factor that could jeopardize participation in the project.

Exclusion Criteria:

* any chronic disease (oncological, cardiovascular, neurological, liver, kidney or other diseases and its acute complications at the discretion of the doctor);
* no cooperation of probands;
* insufficient functional capacity - the presence comorbidities or disorders of the musculoskeletal system, which makes it impossible to complete the training program (assessment by cardiologist, or orthopedist or other specialist);
* smoking, alcohol or drugs abuse;
* non-compliance with epidemiological measures;
* absence of complete vaccination with SARS-CoV-2 vaccine;
* presence of a pacemaker or metal implants (contraindication for magnetic resonance imaging).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximal aerobic capacity | 4 months
  Maximal aerobic capacity parameter of physical fitness will be determined by Rockport walking test (1609m).
Cognitive function testing | 4 months
  All participants will receive extensive psychological testing (Montreal Cognitive Assessment), assessing cognitive domains: attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations, and orientation.
Depressive symptoms | 4 months
  All participants will receive Beck depression questionnaire to identify depressive symptoms.
Olfactory function | 4 months
  The sense of smell will be investigated using the extended "Sniffing' Sticks" test battery, standardized and reliable test used to measure odor thresholds, discrimination & identification.
Brain volumetry (MRI) | 4 months
  Brain MR scans will be performed at 3T PrismaFit scanner using a 64-channel head coil (Siemens Healthcare, Germany).
Molecular genetic analyses | 4 months
  Gene expression will be measured with the aid of qRT-PCR using TaqMan® Gene Expression Assays on the ABI 7900HT (Applied Biosystems, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Ukropcova, Prof., Principal Investigator — Biomedical Research Center Slovak Academy of Sciences
Locations (1):
- Biomedical Research Center Slovak Academy of Sciences, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: 31.12.2025 indefinitely
Access Criteria: In principle to all researchers working in the area. Requests will be reviewed by Prof. Barbara Ukropcova.